CLINICAL TRIAL: NCT02819297
Title: BLI400-302: A Safety and Efficacy Evaluation of BLI400 Laxative in Constipated Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLI400-302
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2020-06-26 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Constipation; Chronic Idiopathic Constipation; CIC
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BLI400 Laxative (Experimental): BLI400 Laxative
  Interventions: Drug: BLI400 Laxative
- Placebo (Placebo Comparator): BLI400 placebo
  Interventions: Drug: BLI400 Placebo

INTERVENTIONS:
Drug: BLI400 Laxative — 21 gm BLI400 powder
  Arms: BLI400 Laxative
Drug: BLI400 Placebo — Equivalent amount of placebo powder
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate a daily dose of BLI400 Laxative for safety and efficacy versus placebo in constipated adults.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years of age
2. Constipated, defined by the following adapted ROME II definition

   Fewer than 3 spontaneous defecations per week and at least one of the following symptoms for at least 12 weeks (which need not be consecutive) in the preceding 12 months:
   * Straining during > 25% of defecations
   * Lumpy or hard stools in > 25% of defecations
   * Sensation of incomplete evacuation for > 25% of defecations
3. If female, and of child-bearing potential, is using an acceptable form of birth control
4. Negative serum pregnancy test at screening, if applicable
5. In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

1. Report loose (mushy) or water stools in the absence of laxative use for more than 25% of BMs during the 12 weeks before Visit 1
2. Meet the Rome II criteria for Irritable Bowel Syndrome.
3. Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon
4. Subjects who have had major surgery 30 days before Visit 1; appendectomy or cholecystectomy 60 days before Visit 1; abdominal, pelvic, or retroperitoneal surgery 6 months before Visit 1; bariatric surgery or surgery to remove a segment of the GI tract at any time before Visit 1
5. Subjects with hypothyroidism that is being treated and for which the dose of thyroid hormone has not been stable for at least 6 weeks at the time of Visit 1
6. Subjects taking laxatives, enemas or prokinetic agents that refuse to discontinue these treatments from Visit 1 until after completion of the study
7. Subjects who are pregnant or lactating, or intend to become pregnant during the study
8. Subjects of childbearing potential who refuse a pregnancy test
9. Subjects who are allergic to any study medication component
10. Subjects taking narcotic analgesics or other medications known to cause constipation
11. Subjects with clinically significant cardiac abnormalities identified at the Visit 1 ECG
12. Subjects with clinically significant laboratory abnormalities, deemed as a potential safety issue by the Investigator
13. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures
14. Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
15. Subjects with an active history of drug or alcohol abuse
16. Subjects have been hospitalized for a psychiatric condition or have made a suicide attempt during the 2 years before Visit 1
17. Subjects who withdraw consent at any time prior to completion of Visit 1 procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories, Inc.
Locations (51):
- United States (51):
  - Braintree Research Site 8, Birmingham, Alabama
  - Braintree Research Site 47, Mobile, Alabama
  - Braintree Research Site 28, Phoenix, Arizona
  - Braintree Research Site 4, Little Rock, Arkansas
  - Braintree Research Site 11, Anaheim, California
  - Braintree Research Site 29, Corona, California
  - Braintree Research Site 35, Garden Grove, California
  - Braintree Research Site 32, La Mirada, California
  - Braintree Research Site 50, Sacramento, California
  - Braintree Research Site 51, Westminster, California
  - Braintree Research Site 36, Denver, Colorado
  - Braintree Research Site 45, Clearwater, Florida
  - Braintree Research Site 10, Hialeah, Florida
  - Braintree Research Site 37, Hialeah, Florida
  - Braintree Research Site 39, Hialeah, Florida
  - Braintree Research Site 2, Miami, Florida
  - Braintree Research Site 6, Miami, Florida
  - Braintree Research Site 38, Miami, Florida
  - Braintree Research Site 52, Miami, Florida
  - Braintree Research Site 19, Miami Lakes, Florida
  - Braintree Research Site 44, Miami Springs, Florida
  - Braintree Research Site 13, Orlando, Florida
  - Braintree Research Site 43, Pembroke Pines, Florida
  - Braintree Research Site 25, Tamarac, Florida
  - Braintree Research Site 3, Tampa, Florida
  - Braintree Research Site 1, West Palm Beach, Florida
  - Braintree Research Site 41, Atlanta, Georgia
  - Braintree Research Site 20, Marietta, Georgia
  - Braintree Research Site 27, Snellville, Georgia
  - Braintree Research Site 46, Meridian, Idaho
  - Braintree Research Site 15, Chicago, Illinois
  - Braintree Research Site 7, Bastrop, Louisiana
  - Braintree Research Site 12, New Orleans, Louisiana
  - Braintree Research Site 24, Las Vegas, Nevada
  - Braintree Research Site 26, Brooklyn, New York
  - Braintree Research Site 17, Hartsdale, New York
  - Braintree Research Site 21, High Point, North Carolina
  - Braintree Research Site 5, Raleigh, North Carolina
  - Braintree Research Site 16, Cincinnati, Ohio
  - Braintree Research Site 30, Cleveland, Ohio
  - Braintree Research Site 48, Columbus, Ohio
  - Braintree Research Site 9, Dayton, Ohio
  - Braintree Research Site 18, Smithfield, Pennsylvania
  - Braintree Research Site 23, Lancaster, South Carolina
  - Braintree Research Site 22, Chattanooga, Tennessee
  - Braintree Research Site 31, Knoxville, Tennessee
  - Braintree Research Site 40, Houston, Texas
  - Braintree Research Site 34, San Antonio, Texas
  - Braintree Research Site 42, West Jordan, Utah
  - Braintree Research Site 14, Newport News, Virginia
  - Braintree Research Site 49, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1020 subjects were consented and entered into a two-week run-in period to confirm constipation status (subjects were required to average < 3 complete spontaneous bowel movements per week). Following the run-in period, 603 subjects qualified for randomization.
Groups:
- BLI400 Laxative: BLI400 Laxative (21 gm of BLI400 powder)
- Placebo: BLI400 placebo (equivalent amount of placebo powder)
Period: Overall Study
Arm/Group | BLI400 Laxative | Placebo
Started | 299 | 304
Completed | 239 | 252
Not Completed | 60 | 52
Not completed — Withdrawal by Subject | 25 | 13
Not completed — Lost to Follow-up | 12 | 14
Not completed — Adverse Event | 12 | 10
Not completed — Physician Decision | 5 | 5
Not completed — Lack of Efficacy | 5 | 8
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- BLI400 Laxative: BLI400 Laxative (21 gm BLI400 powder)
- Total: Total of all reporting groups
Arm/Group | BLI400 Laxative | Placebo | Total
Number analyzed (Participants) | 299 | 304 | 603
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (15.3) | 51.0 (15.9) | 51.7 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 239 | 460
  Male | 78 | 65 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 119 | 114 | 233
  Not Hispanic or Latino | 180 | 190 | 370
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 19 | 21 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 88 | 101 | 189
  White | 187 | 178 | 365
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 299 | 304 | 603

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response
Description: The primary endpoint is the proportion of subjects who are weekly responders for at least 9 out of 12 weeks, with at least 3 of these weeks occurring in the last 4 weeks of treatment. A weekly responder is a subject who has ≥ 3 CSBMs and an increase from baseline of > 1 CSBM in that week.
Time Frame: 12 weeks
Population: modified ITT population - excludes subjects with significant protocol violations
Measure: Count of Participants; unit: Participants
Arm/Group | BLI400 Laxative | Placebo
Number analyzed (Participants) | 294 | 302
Participants | 77 | 39
Statistical Analysis 1: Comparison: BLI400 Laxative vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | BLI400 Laxative | Placebo
All-Cause Mortality (participants affected / at risk) | 0/299 | 0/304
Serious Adverse Events (participants affected / at risk) | 3/299 | 8/304
Other Adverse Events (participants affected / at risk) | 42/299 | 33/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI400 Laxative (N=299) | Placebo (N=304)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI400 Laxative (N=299) | Placebo (N=304)
Flatulence (Gastrointestinal disorders) | 24 (24) | 8 (8)
Urinary tract infection (Infections and infestations) | 20 (20) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT02819297/Prot_SAP_000.pdf